CLINICAL TRIAL: NCT06925854
Title: An Open-label, 2-period, 2-sequence Cross-over Study to Assess the Effect of AZD4144 on the Pharmacokinetics of Rosuvastatin in Healthy Participants
Brief Title: A Study to Investigate How AZD4144 Affects the Pharmacokinetics of Rosuvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D9441C00002
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Nucleotide-binding domain,; leucine-rich-containing family, pyrindomain-containing-3 (NLRP3) inflammasome; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment sequence AB (Experimental): Participants will receive single dose of rosuvastatin under fasted condition (Treatment A), followed by a single dose of rosuvastatin with AZD4144 under fasted condition (Treatment B).
  Interventions: Drug: AZD4144; Drug: Rosuvastatin
- Treatment sequence BA (Experimental): Participants will receive a single dose of rosuvastatin with AZD4144 under fasted condition (Treatment B), followed by a single dose of rosuvastatin under fasted condition (Treatment A).
  Interventions: Drug: AZD4144; Drug: Rosuvastatin

INTERVENTIONS:
Drug: AZD4144 — Oral tablet of AZD4144 will be administered.
Drug: Rosuvastatin — Oral tablet of rosuvastatin will be administered.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of rosuvastatin when administered alone and in combination with single oral dose of AZD4144.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, open label study in healthy participants.

The participants will be provided with:

Treatment A: single dose of rosuvastatin Treatment B: single dose of rosuvastatin in combination with AZD4144. The participants will be randomized in the 1:1 ratio to either receive treatment sequence AB or sequence BA.

The study will be comprised of:

* A screening period of 28 days.
* Two treatment periods (Treatment period 1 and Treatment period 2) of 4 days each where participants will receive the study intervention on Day 1 in Treatment period 1 and on Day 10 in Treatment period 2.
* A final Follow-up visit between Day 17 and Day 20.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index between 18 and 32 kg/m2 inclusive at the Screening Visit and on first admission (Visit 2) to the Clinical Unit and weigh at least 45 kg.
* All females must have a negative pregnancy test at the Screening Visit.
* Female participants of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception.
* Females of non-childbearing potential must be confirmed at the Screening Visit.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods.

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* Clinically significant serious active and chronic infections within 60 days prior to randomisation.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the randomisation.
* Active systemic bacterial, viral, or fungal infection within 14 days prior to dosing or presence of fever (confirmed tympanic body temperature > 37.5 °C) within 14 days prior to dosing on Day 1 depending on experienced symptoms.
* Bacillus Calmette-Guérin vaccine within one year prior to signing the ICF.
* Any laboratory values with deviations at the Screening Visit or on admission to the Clinical Unit. Abnormal values may be repeated at the discretion of the Investigator: alanine transaminase (ALT) >1.00 × Upper Limit Normal (ULN), aspartate transaminase (AST) > 1.00 ×ULN, white blood cell count < Lower limit normal (LLN), differential neutrophils < LLN, bilirubin > 1.00 × ULN, eGlomerular filtration rate (eGFR) < 60 mL/min/1.73 m² calculated using the Chronic Kidney Disease Epidemiology Collaboration equation (eGFR will only be assessed at Screening).
* Any positive result at Screening for serum hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus.
* Has received any investigational medicinal product.
* Participants who have previously received AZD4144.
* Participants with myopathy, defined as muscle weakness that in opinion of the investigator, enhances the participant's risk of developing statin-associated muscle symptoms

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from 0 to infinity (AUCinf) | Day 1 to Day 4 and Day 10 to Day 13
  The AUCinf of rosuvastatin when administered alone and in combination with AZD4144 in healthy participants will be evaluated.
Area under the plasma concentration-curve from 0 to the last quantifiable concentration (AUClast) | Day 1 to Day 4 and Day 10 to Day 13
  The AUClast of rosuvastatin when administered alone and in combination with AZD4144 in healthy participants will be evaluated.
Maximum plasma drug concentration (Cmax) | Day 1 to Day 4 and Day 10 to Day 13
  The Cmax of rosuvastatin when administered alone and in combination with AZD4144 in healthy participants will be evaluated.

SECONDARY OUTCOMES:
Number of participants with adverse events | From screening (Day-28 to Day -2) until Follow-up (Day 20)
  The safety and the tolerability of AZD4144 in combination with rosuvastatin will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure researchenvironmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/